CLINICAL TRIAL: NCT00685334
Title: Atypical Antipsychotic Medication for Outpatients With Anorexia Nervosa
Brief Title: Effectiveness of Atypical Antipsychotic Medication for Outpatients With Anorexia Nervosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4696 (MH069868-01); 1R21MH069868-01 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Eating Disorders
Keywords: Atypical Antipsychotics; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Olanzapine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will take olanzapine
  Interventions: Drug: Olanzapine
- 2 (Active Comparator): Participants will take aripiprazole
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Olanzapine — Participants will take olanzapine daily for 12 weeks.
  Other Names: zyprexa
  Arms: 1
Drug: Aripiprazole — Participants will take aripiprazole daily for 12 weeks.
  Other Names: Abilify
  Arms: 2

SUMMARY:
This study will compare the effectiveness of two atypical antipsychotic medications, olanzapine and aripiprazole, in treating people with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a disease of disordered eating that is characterized by self-starvation, often leading to extreme weight loss and difficulty maintaining a normal weight. Symptoms and behaviors of AN may include distorted body image, obsessive exercise, lack of menstruation among women, binge and purge eating behaviors, and intense fear of weight gain. Furthermore, people with AN are at a high risk of other mental disorders, such as depression and anxiety, and medical complications, such as organ damage, heart failure, and osteoporosis. Current treatments for AN include nutrition counseling, psychotherapy, and medication. Previous studies have suggested that certain medications usually used to treat schizophrenia, also known as atypical antipsychotic drugs, may be helpful in treating people with AN. Specifically, the atypical antipsychotic medications olanzapine and aripiprazole may be effective in improving overall symptoms of AN and in restoring weight to normal levels. This study will compare the effectiveness of olanzapine and aripiprazole in treating people with AN.

Participation in this study will last 12 weeks. All participants will first undergo baseline assessments that will include questionnaires and interviews about AN symptoms, a physical exam, vital sign measurements, an electrocardiograph (EKG), and a blood draw. Participants will then be assigned randomly to 12 weeks of treatment with daily olanzapine or aripiprazole. Participants will meet with a study doctor weekly over the 12 weeks of treatment. During these visits, the study doctor will monitor participants' progress, medication dosage, vital signs, and side effects. In addition, participants will undergo repeat blood draws every 4 weeks and repeat questionnaires every month of the treatment period. Upon completing the 12 weeks of treatment, participants will repeat most baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for AN (DSM-IV criteria for amenorrhea will not be strictly applied, as these patients have been shown to be clinically indistinguishable from those with full criteria AN)
* Body mass index (BMI) less than 19 kg/m2 and greater than 14 kg/m2 (BMI of 19 is equivalent to approximately 85% of ideal body weight [IBW] according to Metropolitan Life standards, and BMI of 14 is equivalent to approximately 65% IBW)
* Unwilling to pursue inpatient treatment if BMI is less than 18 kg/m2
* Free of psychotropic (e.g., antidepressant, antianxiety, mood stabilizer, antipsychotic) medication for 2 weeks before study entry (free for 4 weeks before study entry if taking fluoxetine or antipsychotic medications)
* Prior treatment of AN

Exclusion Criteria:

* Any medical or psychiatric problem requiring urgent clinical attention (e.g., metabolic disturbance, acute suicidality) and/or significant comorbid illnesses that are not likely to benefit from proposed treatments
* Significant orthostatic high blood pressure (systolic change greater than 30 mmHg upon changing from supine to standing position)
* Allergy to olanzapine or aripiprazole
* Commencing psychotherapy in the community within 3 months of study entry
* Diabetes mellitus, with fasting serum glucose greater than 120 mg/dL or nonfasting serum glucose less than 140 mg/dL
* Known history of current or past jaundice
* Known history of narrow angle glaucoma
* Active substance abuse or dependence
* Schizophrenia, schizophreniform disorder, or bipolar illness
* Movement disorder or presence of tics
* History of tardive dyskinesia
* History of seizures
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Attia, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (2):
- New York State Psychiatric Institute, New York, New York, United States
- Toronto General Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine: Dosing of Olanzapine will begin at 2.5 mg and be increased every 2 weeks, first to 5 mg and then 10 mg, if the patient is tolerating the medication. Patients will remain on 10 mg for the final 8 weeks of the trial unless lower doses are necessary.
- Aripiprazole: Aripiprazole dosing will begin at 5 mg daily, and will be increased every two weeks, first to 10 mg daily, then 15 mg daily for the final 8 weeks of the trial, unless lower doses are necessary.
Period: Overall Study
Arm/Group | Olanzapine | Aripiprazole
Started | 12 | 10
Completed | 2 | 3
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 4 | 0
Not completed — Chose to enter hospital | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Aripiprazole | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.7 (7.2) | 30.7 (11.6) | 29.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
  Canada | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight (Lbs.) at 12 Weeks
Description: This study looked at change in weight before and after medication use.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Olanzapine | Aripiprazole
Number analyzed (Participants) | 12 | 10
lbs | 2.2 (6.3) | -1.2 (5.1)

2. Primary Outcome: Tolerability
Description: This study addressed the benefits, tolerability, acceptability, safety, and appropriate dosage of olanzapine and aripiprazole, as determined by clinical evaluation and self report. The outcome measure reported here is the number of patients who did not experience untoward side effects while taking the medication.
Time Frame: Measured at Week 12
Population: Data was not available for all 22 participants.
Measure: Number; unit: Participants
Arm/Group | Olanzapine | Aripiprazole
Number analyzed (Participants) | 8 | 9
Participants | 8 | 9

3. Secondary Outcome: Medication Side Effects
Description: Common side effects include sedation, dizziness, and headache for patients on olanzapine and akathisia, anxiety, dizziness and blurred vision for patients receiving aripriprazole.
Time Frame: Measured at Week 12
Reporting Status: Not Posted
Measure: Number; unit: Participants

4. Secondary Outcome: Treatment Compliance
Description: Total number of randomized patients that completed the full 12 weeks of treatment.
Time Frame: Measured at Week 12
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Arm/Group | Olanzapine | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No